CLINICAL TRIAL: NCT01296373
Title: An Observational Study to Explore Reconstitution of Immunity in Patients With Advanced HIV-1-infection Commencing Combination Antiretroviral Therapy (HIVNAT 136 RESTORE Study:Thailand)
Brief Title: A Study to Explore Reconstitution of Immunity in Patients With Advanced HIV-1-infection
Acronym: RESTORE
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Chulalongkorn University (Other); HIV Netherlands Australia Thailand Research Collaboration (Network); St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: HIVNAT 136
Record Dates: First submitted 2011-02-13; First posted 2011-02-15 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: HIV Immune Restoration
Keywords: HIV-1; immune; restoration; observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, PBMC and DNA will be stored for 10 years total.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1-infected, off ART: HIV-1-infected, antiretroviral naive or off antiretroviral therapy for at least 12 months with CD4+ T-cell counts less than or equal to 350 cells/µL who are about to commence combination antiretroviral therapy

SUMMARY:
RESTORE study:Thailand is a prospective observational study of HIV-1-infected patients who are either treatment naïve or who have been off anti-retroviral therapy for a ≥12 months, who have a CD4+ T cell count less than or equal to 350 cells/µL and who have been deemed by their treating physician that commencement of combination antiretroviral therapy (cART), which is expected to reduce plasma HIV RNA by ≥1log10 copies/mL, is necessary.

The primary intent of this protocol is to prospectively establish a cohort of patients from whom clinical data and peripheral blood samples (serum, plasma and peripheral blood mononuclear cells) can be stored for substudies examining reconstitution of the immune system and its relationship to disease outcomes.

DETAILED DESCRIPTION:
RESTORE study:Thailand is a prospective observational study of HIV-1-infected patients who are either treatment naïve or who have been off anti-retroviral therapy for a ≥12 months, who have a CD4+ T cell count less than or equal to 350 cells/µL and who have been deemed by their treating physician that commencement of combination antiretroviral therapy (cART) which is expected to reduce plasma HIV RNA by ≥1log10 copies/mL is necessary.

The primary intent of this protocol is to prospectively establish a cohort of patients from whom clinical data and peripheral blood samples (serum, plasma and peripheral blood mononuclear cells) can be stored for substudies examining reconstitution of the immune system and its relationship to disease outcomes.

Patients who have recently had an opportunistic infection (OI) can also be enrolled. Investigators should consider the results of the ACTG A5164 (1), SAPIT (2), and Makadzange and colleagues (3) studies in regard to the timing of cART introduction following the acute OI. This observational protocol does not stipulate the timing of cART introduction, but cART should not normally be delayed beyond 2 months after the diagnosis of an acute OI.

Patients will be commenced on cART regimens as determined by the treating physician. Patients will be observed and pertinent clinical data will be recorded at visits that will coincide with their standard of care visits. The visit schedule in year 1 is as follows: screening/baseline (cART is commenced), week 4, 8, 12, 24 and 48. In year 2 and 3 visits are every 6 months. In those who, in the opinion of the investigator, develop a major clinical manifestation of immune restoration disease (IRD) an extra visit (IRD baseline) will be conducted. If the patient is in the first 12 weeks of study follow-up, this is the only additional visit required. If, however, the major IRD event occurs after the week 12 visit in year 1 or in years 2 and 3, in addition to the IRD baseline visit a second additional visit will be conducted 4 weeks later. It is likely that these extra visits would be required for the management of their clinical disease. Details pertaining to the cause, course and treatment of the IRD event will be recorded. These will include clinical data and pathology results. Prior to starting cART and at each study visit, extra blood samples will be taken for storage and subsequent analysis. It is envisaged that these storage samples will be used for subsequent exploration of aspects of immunity (including but not limited to pathogen specific immune responses including pathogen load; anti-HIV immunity; pathogen specific (and other) clinical syndromes associated with immune reconstitution; B-cell responses); immune activation and HIV viral dynamics. A sample for genetic testing will be obtained at baseline. The rationale for this is to determine host genetic polymorphisms that may predict immune reconstitution with cART and/or predispose to the development of IRD. Patients will be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

. Age ≥18 years;

* Provision of written, informed consent;
* Untreated, HIV infected patients with CD4+ T cell counts 350 cells/µL or less;
* Treatment naïve or off ART for ≥12 months;
* Intention to commence cART that would be expected to reduce viral load by one log or greater

Exclusion Criteria:

* Inability to give written informed consent;
* Any condition which the treating physician feels would compromise the ability of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected adults aged 18 years or older with untreated HIV-1-infection and CD4+ of 350 cells/uL or less who are about to start or recommence combination antiretroviral therapy which is expected to result in a 1 log or greater decline in plasma HIV RNA
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Longitudnal Changes in CD4+ T-cell with combination antiretoviral therapy | 2-3 years

SECONDARY OUTCOMES:
Longitudinal changes in T-cell subsets with combination antiretroviral therapy | 2-3 years
Longitudinal changes in CD4+ T-cell immune responses to common pathogens during combination antiretroviral therapy | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Pett, MD, Study Director — National Centre in HIV Epidemiology and Clinical Research.; David A Cooper, MD, Study Chair — National Centre in HIV Epidemiology and Clinical Research.; Anthony D Kelleher, MD, Study Chair — St Vincent's Hospital, Sydney; Denise Hsu, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Jintanat Ananworanich, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- [Derived] Hsu DC, Kerr SJ, Iampornsin T, Pett SL, Avihingsanon A, Thongpaeng P, Zaunders JJ, Ubolyam S, Ananworanich J, Kelleher AD, Cooper DA. Restoration of CMV-specific-CD4 T cells with ART occurs early and is greater in those with more advanced immunodeficiency. PLoS One. 2013 Oct 10;8(10):e77479. doi: 10.1371/journal.pone.0077479. eCollection 2013. PMID 24130889